CLINICAL TRIAL: NCT04975724
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Clinical Trial to Assess Safety and Effectiveness of Liposom in Enhance and Speed up Response With Citalopram in Elderly Patients Suffering From Major Depressive Disorder (MDD)
Brief Title: Safety of Liposom With Citalopram in Elderly Patients With Major Depressive Disorder
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fidia Farmaceutici s.p.a. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QQ05.16.02
Record Dates: First submitted 2020-03-02; First posted 2021-07-23 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — liposom; Citalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A Liposom Forte + Citalopram (Experimental): Liposom Forte (2 ampoules of 28mg/2 ml) for 30 days + citalopram (10mg) for 90 days
  Interventions: Drug: Liposom Forte; Drug: Citalopram
- Group B Placebo + Citalopram (Experimental): Placebo (2 ampoules of 2 ml) for 30 days + citalopram (10mg) for 90 days
  Interventions: Drug: Citalopram; Other: Placebo

INTERVENTIONS:
Drug: Liposom Forte — Liposom Forte 28mg/2ml solution for injection contains a mixture of purified hypothalamic phospholipids (PLs) from swine brains. The key components of the phospholipid mixture are phosphatidylcholine (PC), phosphatidylethanolamine (PE) and phosphatidylserine (PS).
  Other Names: Liposom
  Arms: Group A Liposom Forte + Citalopram
Drug: Citalopram — The medicinal product Citalopram Aurobindo contains citalopram as active ingredient available on the market in 20 mg film coated tablets. The tablets are divisible in two equal part of 10 mg as reported in the SmPC
Other: Placebo — Liposom Forte Placebo (2 ampoules of 2 ml solution for injection)
  Other Names: Placebo of Liposom Forte
  Arms: Group B Placebo + Citalopram

SUMMARY:
The purpose of this study is to determine if Liposom Forte will enhance the response to antidepressant therapy with citalopram in elderly patients suffering from Major Depressive Disorder (MDD).

DETAILED DESCRIPTION:
The effects of phospholipid liposomes when associated with antidepressant drugs are very interesting. In addition to an improvement of somatic symptoms of depression, measured with the Hamilton Rate Scale for Depression, liposomes are able to reduce the latency of onset of the antidepressant activity of drugs like amitriptyline, clomipramine, and trazodone. These results indicate that phospholipids can be used as an adjuvant to antidepressant therapy, also allowing specific antidepressant drug dose reduction. Thus, the hypothesis is that combination therapy would not only lead to greater efficacy, but also to a more rapid onset of therapeutic response. The addition of Liposom Forte may be clinically important since it may ensure the use of lower citalopram doses, thereby reducing the risk of adverse events, and this may prove to be important, especially in elderly people.

ELIGIBILITY:
Inclusion Criteria:

1. Meets DSM-V criteria for major depressive disorder
2. Score of ≥ 16 in the HAM-D
3. Score of ≥ 23 on the Mini-Mental State Exam (MMSE-2)
4. Aged ≥ 65 and < 85 years
5. Patients able to understand the study procedures and to comply with protocol requirements
6. Patients legally able to give written informed consent to the trial (signed and dated by the subject)

Exclusion Criteria:

1. Any contraindication for treatment or intolerance to Liposom Forte or citalopram
2. Congenital long QT syndrome, bradycardia, recent acute myocardial infarction, uncompensated heart failure or concomitant use of drugs that prolong the QT interval
3. History of psychiatric disorder other than major depressive disorder, including history of substance use disorder
4. Presence of psychotic symptoms, even if they are not sufficient to make diagnosis of a mental disorder
5. Severe organic disease (e.g., major surgery, metastatic cancer, stroke, delirium, severe neurological disorder, heart attack, chronic heart failure, asthma, severe cardio circulatory disorders)
6. Diabetes Mellitus type I and II
7. Acute suicidal or violent behaviour or history of suicide attempt within the year prior to study entry or current suicidal ideation
8. Treated with long acting injectable (LAI) antipsychotics within 6 months prior to study entry
9. Treated with any antipsychotics, antidepressant, food supplements or over-the-counter CNS-active medications (e.g, St. John's Wort, melatonin, Selective Serotonin Reuptake Inhibitors [SSRIs], Serotonin and norepinephrine reuptake inhibitors [SNRIs], Monoamine-Oxidase Inhibitors [MAOIs], or other antidepressants) within 4 weeks prior to the first administration of study medication
10. Ongoing or planned psychotherapy or other psychological treatment during the study period

Ages: 65 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-04-18 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change of depressive symptoms atV5(day30)as change from baseline with HamiltonRatingScaleforDepression (21items,scoring based on the first17.9items from0=not present;to4=severe.8 from0-2.Scores from the first17items summed:≥16=MajorDep) | Day 30 (V5)
  The purpose of this study is to determine if Liposom Forte will enhance the response to antidepressant therapy with citalopram in elderly patients suffering from Major Depressive Disorder (MDD). HamiltonRatingScaleforDepression (21items,scoring based on the first17.9items from0=not present;to4=severe.8 from0-2.Scores from the first17items summed:≥16=MajorDep)

SECONDARY OUTCOMES:
Change of latency of antidepressant therapy with citalopram. Evaluated at V2,V3,V4 and V5 using HamiltonRatingScaleforDepression Latency time:the time from baseline to response (a≥50% improvement in HAM-D score vs baseline) | From baseline through 30 days follow-up (V5)
  Determine if Liposom Forte will speed up response to antidepressant therapy with citalopram HamiltonRatingScaleforDepression (21items,scoring based on the first17.9items from0=not present;to4=severe.8 from0-2.Scores from the first17items summed:≥16=MajorDep)
ClinicalGlobalImpression as change from baseline up toV8Day90.CGI:7point scale clinician-rated(severity of illness)from1(normal)to7(severely ill).CGI score from1(very much improved)to7(very much worse).Treatment response consider efficacy andAEs | From baseline through 90 days follow-up (V8)
  Determine the Clinical Global Impression to treatments
Safety of study treatments by tracking number and type of adverse events at each visit, up to V8 (Day 90) | From baseline through 90 days follow-up (V8)
  To assess the safety of study treatments
Safety of study treatments by tracking, up to V8 (Day 90), 12-lead ECG, QTcF interval (Fridericia equation) will be measured | From baseline to Day 14 (V3) and Day 90 (V8)
  To assess the safety of study treatments
Safety of study treatments by tracking, up to V8 (Day 90), blood pressure measurements in mmHg | From baseline through 90 days follow-up (V8)
  To assess the safety of study treatments tracking blood pressure measurement in mmHg
Safety of study treatments by tracking, up to V8 (Day 90), heart rate measurements in bpm | From baseline through 90 days follow-up (V8)
  To assess the safety of study treatments tracking heart rate
Safety of study treatments by tracking, up to V8 (Day 90), oxygen saturation measurements in percentage with a pulse oximetry device | From baseline through 90 days follow-up (V8)
  To assess the safety of study treatments tracking oxygen saturation
Change of depressive symptoms during the entire study as change from baseline therapy with citalopram over the entire study | From baseline through 90 days follow-up (V8)
  Change of depressive symptoms will be evaluated over the entire study as change from baseline using the HAM-D (Hamilton Rating Scale for Depression). The score is based on the first 17 items: nine items are scored on a 5-point scale, ranging from 0 = not present to 4 = severe. Eight are scored from 0-2. The score is summed and patients are categorized as follows: 0-7 = No depression 8-15 = Minor Depression
  ≥ 16 = Major Depression
Percentage of patients responders at V2, V3, V4 and V5. ≥50% improvement in HAM-D score vs baseline will be considered as responder. | From baseline through 30 days follow-up (V5)
  determine if Liposom Forte will speed up response to antidepressant therapy with citalopram
Change of depressive symptoms as change from baseline using Geriatric Depression Scale (GDS-15). | From baseline through 90 days follow-up (V8)
  Change of depressive symptoms will be evaluated over the entire study. GDS:brief questionnaire:15questions with options yes or no in reference to how patients felt on the day of administration. Answers indicating depression are in bold and italicized; score one point for each one selected. A score of 0 to 5 is normal. A score greater than 5 suggests depression.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Giordan, Study Director — Fidia Farmaceutici s.p.a.
Locations (12):
- Italy (12):
  - UOC Geriatria e Lungodegenza Geriatrica PO San Filippo e Nicola di Avezzano - ASL1 Avezzano Sulmona L'aquila, Avezzano
  - UO Psichiatria - ASST Papa Giovanni XXIII, Bergamo
  - Ambulatorio Psichiatrico, UOC Psichiatria Presidio Ospedaliero di Codogno - ASST Lodi, Codogno
  - SOD Geriatria-UTIG Azienda Ospedaliero-Universitaria Careggi, Florence
  - Servizio Psichiatrico di Diagnosi e Cura (SPDC) Foggia, Ospedali Riuniti di Foggia, Foggia
  - Servizio Psichiatrico di Diagnosi e Cura (SPDC) - ASL3 Ente Ospedaliero Ospedali Galliera, Genova
  - Ambulatorio Clinica Psichiatrica, Ospedale Policlinico S. Martino, Genova
  - UOC Geriatria PO San Salvatore - ASL1 Avezzano Sulmona L'Aquila, L’Aquila
  - SPDC Ospedale Fatebenefratell, UOC Psichiatria 1 ASST Fatebenefratelli Sacco, Milan
  - Centro Depressione Anziani S.C. Psichiatria 51, ASST Santi Paolo e Carlo - Presidio San Paolo, Milan
  - UOC Psichiatria - Azienda Ospedaliero-Universitaria Sant'Andrea, Roma
  - Clinica Psichiatrica, Azienda Sanitaria Universitaria Integrata di Udine, Udine